CLINICAL TRIAL: NCT03446690
Title: The Use of MI Varnish for the Prevention and Reduction of White Spot Lesions in Orthodontic Treatment
Brief Title: MI Varnish for the Prevention of White Spot Lesions
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Alabama at Birmingham (Other)
Responsible Party: Principal Investigator, Chung How Kau, Professor and Chairman, University of Alabama at Birmingham
Allocation: Non-Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 1135815
Record Dates: First submitted 2018-02-14; First posted 2018-02-27 (Actual); Results first posted 2018-06-12 (Actual); Last update posted 2023-06-26 (Actual); Status verified 2023-06

CONDITIONS: White Spot Lesion; Orthodontic Treatment
Keywords: Enamel decalcification
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: 33 subjects were prospectively recruited for the project in the MI Varnish group. These subjects were studied against a control group of 29 orthodontically treated subjects who received routine treatment and oral hygiene regimes. All subjects will be patients seeking orthodontic treatment at the Department of Orthodontics, School of Dentistry, University of Alabama at Birmingham.
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- MI Varnish Group (Experimental): 33 subjects were prospectively recruited for the project in the MI Varnish group. All subjects will be patients seeking orthodontic treatment at the Department of Orthodontics, UAB. MI Varnish were applied on their teeth initially for 4 weeks (twice) and then 3 monthly intervals.
  Interventions: Drug: MI Varnish
- Control group (Other): A control group was comprised of 29 orthodontically treated subjects who received routine treatment and oral hygiene regimes. All subjects will be patients seeking orthodontic treatment at the Department of Orthodontics, School of Dentistry, University of Alabama at Birmingham. No intervention for this group.
  Interventions: Other: Control group

INTERVENTIONS:
Drug: MI Varnish — MI Varnish with RECALDENT™ (CPP-ACP) enhances enamel acid resistance and boosts salivary fluoride levels. This product remains on the teeth longer than other fluoride varnishes and contains high levels of fluoride and calcium released in the oral cavity. The difference is in the RECALDENT™ (CPP-ACP), which makes MI Varnish a natural and unique choice for your patients. Casein phosphopeptides (CPP) naturally occurs in milk casein; Amorphous Calcium Phosphate (ACP), which is found in the RECALDENT™, is also the source of calcium and phosphate. In the oral cavity, CPP binds to oral surfaces such as teeth, dentin, oral mucosa and biofilm. Calcium and phosphate ions are the building blocks for healthy teeth and MI Varnish delivers bioavailable calcium and phosphate ions into the saliva.
  Arms: MI Varnish Group
Other: Control group — Participants received routine treatment and oral hygiene regimes. No intervention for this group.
  Arms: Control group

SUMMARY:
The current study aimed to determine if MI Varnish has an effect in preventing the formation of white spot lesions for patients undergoing orthodontic treatment. 33 subjects were prospectively recruited for the project as the MI Varnish group, with a control group of 29 orthodontically treated subjects who received routine treatment and oral hygiene regimes.Difference in prevention of white spot formation between the control and the study groups were evaluated through photographic records and clinical examination by using the Enamel Decalcification Index (EDI) scores.

DETAILED DESCRIPTION:
Orthodontists face two common iatrogenic treatment side effects, root resorption and enamel decalcification, with the latter occurring at a much higher frequency. While the processes that lead to enamel demineralization are understood, methods to diminish or perhaps eliminate degradation of enamel surfaces are being searched for. A new product, MI Varnish, is current available and has been shown in some initial case reports to be useful in reducing white spot lesions. It contains a special milk-derived protein RECALDENT TM (CPP-ACP) in which the casein phosphopeptides (CPP) bind to teeth, dentin, and oral mucosa while the amorphous calcium phosphate (ACP) releases calcium and phosphate. The current study aimed to determine if MI Varnish has an effect in preventing the formation of white spot lesions for patients undergoing orthodontic treatment. 33 subjects were prospectively recruited for the project as the MI Varnish group, with a control group of 29 orthodontically treated subjects who received routine treatment and oral hygiene regimes. The study group received the MI Varnish on the day of bracket bonding. Subjects were recalled initially for 4 weeks (twice) and then at 3 monthly intervals. Difference in prevention of white spot formation between the control and the study groups were evaluated through photographic records and clinical examination by using the Enamel Decalcification Index (EDI) scores.

ELIGIBILITY:
Inclusion Criteria:

* Patients seeking orthodontic treatment and receiving routine treatment and oral hygiene regimes.

Exclusion Criteria:

* Any medical or dental condition that in the opinion of the investigator could impact study results during the expected length of the study;
* Patient is currently using any investigational drug or any other investigational device;
* Patient plans to relocate or move within six months of enrollment.

Ages: 10 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 62 (Actual)
Dates: Start 2015-01-01 (Actual); Primary Completion 2015-11-01 (Actual); Study Completion 2016-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Chung H Kau, BDS, PhD, Principal Investigator — University of Alabama at Birmingham

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Groups:
- MI Varnish Group: 33 subjects were initially recruited in the study for MI Varnish. 7 subjects failed to return or did not meet the study protocol. 29 subjects were recruited retrospectively from a previous study and the results compared.
  MI Varnish were applied on their teeth initially for 4 weeks (twice) and then 3 monthly intervals.
- Control Group: A control group was comprised of 29 orthodontically treated subjects who received routine treatment and oral hygiene regimes. No intervention for this group.
  Control group: Participants received routine treatment and oral hygiene regimes. No intervention for this group.
Period: Overall Study
Arm/Group | MI Varnish Group | Control Group
Started | 33 | 29
Completed | 26 | 29
Not Completed | 7 | 0

BASELINE CHARACTERISTICS:
Groups:
- MI Varnish Group: 33 subjects were prospectively recruited for the project in the MI Varnish group. All subjects will be patients seeking orthodontic treatment at the Department of Orthodontics, UAB.
- Control Group: A control group was comprised of 29 orthodontically treated subjects who received routine treatment and oral hygiene regimes. All subjects were patients seeking orthodontic treatment at the Department of Orthodontics, School of Dentistry, University of Alabama at Birmingham.
- Total: Total of all reporting groups
Arm/Group | MI Varnish Group | Control Group | Total
Number analyzed (Participants) | 26 | 29 | 55
Age, Continuous [Mean (Standard Deviation); unit: years] | 29.5 (6.7) | 28.5 (5.2) | 29 (5.94)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16 | 16 | 32
  Male | 10 | 13 | 23
Region of Enrollment [Count of Participants; unit: Participants]
  Central America | 18 | 20 | 38
  Africa | 6 | 9 | 15
  China | 2 | 0 | 2

OUTCOME MEASURES:

1. Primary Outcome: Enamel Decalcification Index (EDI) Scores
Description: Photographic records will be used to determine the improvements in the white spot lesions. A standard intra-oral photographic camera will be utilized and the photographs will be taken in a light controlled environment and photographs will be captured in a pre-set photographic protocol. The Enamel decalcification index (EDI) will be used to determine the number of white spot lesions present at each time frame.Enamel decalcification index calculation: The facial surface of each tooth was divided into 4 areas (m, Mesial; g, gingival; d, distal; o, occlusal). A score was allocated for each area of each tooth: 0, no decalcification, to 3, decalcifications covering 100% of the area at each time period. Analysis was done at the tooth level, aggregating the enamel decalcification scores from all four areas, creating an EDI for each tooth ranging potentially from 0 to 12. Higher EDI scores indicate more decalcification of teeth and represent a worse outcome.
Time Frame: Photographs were taken for 4 times at monthly intervals. EDI scores were measured and assessed at 1, 2, 3 and 4 months, Month 4 reported. The duration of the observation is an average of 4 months.
Measure: Mean (95% Confidence Interval); unit: scores on a scale
Groups:
- MI Varnish Group: 33 subjects were initially recruited in the study for MI Varnish. 7 subjects failed to return or did not meet the study protocol. MI Varnish were applied on their teeth initially for 4 weeks (twice) and then 3 monthly intervals.
Arm/Group | MI Varnish Group | Control Group
Number analyzed (Participants) | 26 | 29
scores on a scale
  Total EDI score of 1-month visit | 1.038 [0.268 to 1.809] | 1 [0.382 to 1.618]
  Total EDI score of 2-month visit | 1.308 [0.138 to 2.477] | 2.724 [0.769 to 4.679]
  Total EDI score of 3-month visit | 1.923 [0.382 to 3.464] | 3.966 [1.662 to 6.269]
  Total EDI score of 4-month visit | 2.692 [0.778 to 4.607] | 5.897 [3.028 to 8.765]

ADVERSE EVENTS:
Time Frame: During and within 6 months from the end of the treatment.
Arm/Group | MI Varnish Group | Control Group
All-Cause Mortality (participants affected / at risk) | 0/33 | 0/29
Serious Adverse Events (participants affected / at risk) | 0/33 | 0/29
Other Adverse Events (participants affected / at risk) | 0/33 | 0/29

LIMITATIONS AND CAVEATS:
We attempt to overcome the compliance barrier giving the patients brushing technique instructions as a control of their actual compliance with the protocol. However it was observed plaque accumulation and gingival inflammation on some patients.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less

DOCUMENTS (2):
  • Study Protocol (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03446690/Prot_000.pdf
  • Statistical Analysis Plan (2018-01-01): https://cdn.clinicaltrials.gov/large-docs/90/NCT03446690/SAP_001.pdf